CLINICAL TRIAL: NCT03123211
Title: Expanded Access to Veliparib
Status: No longer available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C16-468; C19-918 (Other Grant/Funding Number: AbbVie); C20-120 (Other Grant/Funding Number: AbbVie)
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Solid Tumors With Documented BRCA, BARD, or PALB or Other Acceptable DNA Mutations or Anomalies That Are Scientifically Sound; Triple Negative Breast Cancer (TNBC); High Grade Serous Ovarian Cancer; Patients Requiring Veliparib Suspension Formulation
Keywords: Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — veliparib

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate

INTERVENTIONS:
Drug: Veliparib — Veliparib will be administered orally.
  Other Names: ABT-888

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to veliparib prior to approval by the local regulatory agency. Availability will depend on territory eligibility. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria. EAP is also available for other indications where there is reasonable scientific basis for efficacy.

DETAILED DESCRIPTION:
Expanded Access

ELIGIBILITY:
Inclusion Criteria:

* The patient has relapsed/refractory disease and exhausted all standard treatments.
* The patient has documented Breast Cancer (BRCA), BRCA associated RING domain (BARD), or Partner and Localizer of Breast Cancer (PALB) or other acceptable deoxyribonucleic acid (DNA) mutations.

Exclusion Criteria:

* The patient is eligible for a Poly Adenosine diphosphate ribose polymerase (PARP) inhibitor clinical trial.
* The patient has previously received a PARP inhibitor for the same disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie